CLINICAL TRIAL: NCT04062799
Title: Identification of an Immunophenotype of Risk of Poor Prognosis in Elderly Patients Who Have Been Admitted for Pneumonia
Brief Title: Immunophenotype of Risk in Older Patients Admitted for Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-NEU-2018-118
Record Dates: First submitted 2019-05-06; First posted 2019-08-20 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Age Associated Immune Deficiency; Elderly Infection; Pneumonia; Nutrition Disorders in Old Age; Frail Elderly Syndrome; Sarcopenia
MeSH Terms: conditions — Pneumonia; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — It is an observationa study. There is no intervention.

SUMMARY:
The objective is to evaluate if the immune risk phenotype (IRP) in patients who have been admitted for pneumonia predisposes to worse long-term outcomes. In addition, the association between the detected immunological alterations and clinical, functional, nutritional or comorbidity risk factors will be evaluated.

If the hypothesis is confirmed, helpful immunological markers will be identified. This will be useful in clinical practice to identify patients who can benefit from an intervention and / or to identify the best time for vaccination. Otherwise, valuable information will be obtained on the interrelation between immunological, clinical, functional and nutritional aspects.

DETAILED DESCRIPTION:
The objective is to evaluate if the immune risk phenotype (IRP) in patients who have been admitted for pneumonia predisposes to worse long-term outcomes. In addition, the association between the detected immunological alterations and clinical, functional, nutritional or comorbidity risk factors will be evaluated.

Methodology: Prospective observational study. It will include 149 patients ≥ 65 years admitted for pneumonia. After 30-45 days of pneumonia diagnosis, a complete clinical, functional, nutritional and immunological assessment will be carried out. FRI will be defined as a positive cytomegalovirus serology together with at least one of the following: CD4 / CD8 <1, CD8 T cells> 600 / μl or negative CD28 T cells> 300 / μl15. Mortality and re-admissions at 12 and 18 months will be evaluated.

If the hypothesis is confirmed, helpful immunological markers will be identified. This will be useful in clinical practice to identify patients who can benefit from an intervention and / or to identify the best time for vaccination. Otherwise, valuable information will be obtained on the interrelation between immunological, clinical, functional and nutritional aspects.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 65 years old admitted for pneumonia in the "Hospital de la Santa Creu i Sant Pau in Barcelona".

Exclusion Criteria:

* patients from another acute care hospital
* patients with HIV infection
* neutropenic patients (neutrophil count <1000 / mm3)
* transplant patients
* patients in end-of-life situation
* not having written informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥ 65 years old admitted for pneumonia in the "Hospital de la Santa Creu i Sant Pau in Barcelona".
  Pneumonia will be defined in the presence of a new infiltrate in the chest radiograph along with one or more compatible signs or symptoms: fever, chills, cough, expectoration or malaise.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Presence of the immune risk phenotype (IRP) | 18 months
  To assess whether the presence of the immune risk phenotype (IRP) in patients who have been admitted for pneumonia predisposes to higher mortality after 18 months of pneumonia.

SECONDARY OUTCOMES:
Number of readmissions | 18 months
  To assess number of readmissions at 18 months.
Immunological markers other than IRP | 18 months
  To evaluate if immunological markers other than IRP predispose to higher mortality or readmission rates
Immunological profile | 18 months
  To describe the basic immunological profile of the elderly who have been admitted due to pneumonia and its evolution after the acute phase.
Immunological alterations | 18 months
  To study if there is an association between IRP and clinical, functional, nutritional, comorbidity risk factors or frailty/sarcopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Olga H Torres, PhD MD, Principal Investigator — Hospital de Sant Pau. Universitat Autònoma de Barcelona. Institut de Recerca Sant Pau.
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided